CLINICAL TRIAL: NCT03988413
Title: Single-center, Randomized, Double-blind, Placebo-controlled, Single Dose Ascending Trial of SYHA1402 Tablets in Healthy Subjects
Brief Title: Study on Safety, Absorption and Metabolism of SYHA1402 Tablets in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYHA1402201801/PRO-1
Record Dates: First submitted 2019-06-10; First posted 2019-06-17 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2019-06

CONDITIONS: Diabetic Neuropathy Peripheral
MeSH Terms: interventions — Magnesium-25

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 25mg (Experimental): Tablets, Oral, 25mg, single dose
  Interventions: Drug: 25mg
- 50mg (Experimental): Tablets, Oral, 50mg, single dose
  Interventions: Drug: 50mg
- 100mg (Experimental): Tablets, Oral, 100mg, single dose
  Interventions: Drug: 100mg
- 200mg (Experimental): Tablets, Oral, 200mg, single dose
  Interventions: Drug: 200mg
- 400mg (Experimental): Tablets, Oral, 400mg, single dose
  Interventions: Drug: 400mg
- 800mg (Experimental): Tablets, Oral, 800mg, single dose
  Interventions: Drug: 800mg

INTERVENTIONS:
Drug: 25mg — SYHA1402 25mg or Placebo 25mg
  Arms: 25mg
Drug: 50mg — SYHA1402 50mg or Placebo 50mg
  Arms: 50mg
Drug: 100mg — SYHA1402 100mg or Placebo 100mg
  Arms: 100mg
Drug: 200mg — SYHA1402 200mg or Placebo 200mg
  Arms: 200mg
Drug: 400mg — SYHA1402 400mg or Placebo 400mg
  Arms: 400mg
Drug: 800mg — SYHA1402 800mg or Placebo 800mg
  Arms: 800mg

SUMMARY:
The trial used single-center, randomized, double-blind, placebo-controlled, single-dose study.

The trial planned to enroll sixty-two healthy volunteers. The subjects were allocated to seven dose groups, including 25 mg (4+2), 50 mg (8+2), 100 mg (8+2), 200 mg (8+2), 400 mg (8+2), 800 mg (6+2) and 1200 mg (6+2). Each dose group was allocated test drugs and placebos according to the proportion of subjects in the brackets mentioned above.

ELIGIBILITY:
Inclusion Criteria:

1. 18≤Age≤45, male or female;
2. Body weight (> 45.0 kg (female) or 50.0 kg (male), 19.0 kg/m2 (< BMI) = 26.0 kg/m2);
3. Subjects with normal clinical significance by medical history, vital signs, physical examination and laboratory examination;
4. All subjects who adopt effective non-hormonal contraceptive measures (such as condoms, intrauterine devices without drugs, etc.) from the signing of informed consent to three months after the end of the study;
5. Subjects who voluntarily signed the informed consent and are able to cooperate to complete the test according to the protocal.

Exclusion Criteria:

1. Female subjects: pregnant or lactating, or planned pregnancy; male subjects: their partner planned pregnancy, or planned to donate sperm;
2. Have neurological or psychiatric diseases history, or have serious cardiovascular, liver and kidney, endocrine, respiratory, blood, digestive, immune and other systemic diseases history;
3. Surgery history within six months before signing the informed consent;
4. Allergic history to more than one drug or other serious allergic rhistory.
5. Subjects with a QTc interval greater than 450 ms (male) or 470 MS (female), or with a history of prolonged QTc interval;
6. Positive with serum immunological test for HBsAg, Anti-HCV, Anti-HIV or Anti-TP;
7. History of drugs or drug abuse or alcoholics;
8. History of blood donation more than 200 mL within 8 weeks before signing informed consent;
9. Subjects participating in other clinical trials, or who have participated in any other clinical trials of drugs within three months before signing informed consent;
10. Not suitable for this trial according to the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Change of systolic blood pressure and diastolic blood pressure | 0, 0.5, 1, 2, 4, 8, 12, 24, 48, 72 hours
  To assess the change of blood pressure after administration of SYHA1402
Change of heart rate | 0, 0.5, 1, 2, 4, 8, 12, 24, 48, 72 hours
  To assess the change of heart rate after administration of SYHA1402
Change of pulse | 0, 0.5, 1, 2, 4, 8, 12, 24, 48, 72 hours
  To assess pulse after administration of SYHA1402
Change of body temperature | 0, 0.5, 1, 2, 4, 8, 12, 24, 48, 72 hours
  To assess the change of body temperature after administration of SYHA1402
Change of 12-lead ECG | 0, 0.5, 1, 2, 4, 8, 24, 48, 72 hours
  To assess the change of 12-lead ECG (PR，QRS，QT，QTc) after administration of SYHA1402
Change of physical examination | 24, 48, 72 hours
  To assess the change of physical examination (including cardiovascular system, chest and lung, abdomen, nervous system, skeletal muscle system, etc) after administration of SYHA1402
Change of blood biochemistry | 24, 48, 72 hours
  To assess the change of blood biochemistry (including LDL, HDL,TC, ALT, AST, etc) after administration of SYHA1402
Chagne of blood routine | 24, 48, 72 hours
  To assess the change of blood routine after administration of SYHA1402
Change of urinary routine | 24, 48, 72 hours
  To assess the change of urinary routine after administration of SYHA1402

SECONDARY OUTCOMES:
Peak concentration (Cmax) | 10minutes, 20minutes, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72 hours
  Plasma peak concentration (Cmax) after administration of SYHA1402
Peak time (Tmax) | 10minutes, 20minutes, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72 hours
  Plasma peak time (Tmax) after administration of SYHA1402
Area under the plasma concentration-time curve (AUC0-72h) | 10minutes, 20minutes, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72 hours
  The area under the plasma concentration-time curve of SYHA1402 after administration are calculated.
Half time (t1/2) | 10minutes, 20minutes, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72 hours
  The half time of SYHA1402 after administration are calculated.
Apparent clearance (CL/F) | 10minutes, 20minutes, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72 hours
  To assess the apparent clearance (CL/F) after administration of SYHA1402
Proportional dose-response relationship between pharmacokinetic parameters Cmax and AUC of SYHA1402 | 10minutes, 20minutes, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72 hours
  To assess the Proportional dose-response relationship between pharmacokinetic parameters Cmax and AUC of SYHA1402

CONTACTS AND LOCATIONS:
Locations (1):
- The General Hospital of the People's Liberation Army, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liang B, Wang J, Zhang G, Wang R, Cai Y. Safety, Tolerability and Pharmacokinetics of Single-Dose Oral SYHA1402 in Healthy Chinese Subjects. Neurol Ther. 2023 Jun;12(3):947-959. doi: 10.1007/s40120-023-00480-x. Epub 2023 Apr 24. PMID 37093466